CLINICAL TRIAL: NCT02947607
Title: Investigation of the Role of the Microbiome in the Pathogenesis of Colorectal Adenoma and Carcinoma
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry); KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s57084
Record Dates: First submitted 2016-10-13; First posted 2016-10-28 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Adenoma and Carcinoma
Keywords: Human gut microbiome; Colorectal cancer; Colorectal adenoma; Gut bacteria; Metagenomics; Metatranscriptomics
MeSH Terms: conditions — Carcinoma; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Stool Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy control: Patients undergoing lower GI endoscopy without any colorectal adenoma or carcinoma.
  Interventions: Procedure: Colon biopsies
- Adenoma: Patients undergoing lower GI endoscopy with presence of colorectal adenoma detected.
  Interventions: Procedure: Colon biopsies
- Colorectal cancer: Patients diagnosed with colorectal cancer and referred to surgical carcinoma resection.
  Interventions: Procedure: Colon biopsies

INTERVENTIONS:
Procedure: Colon biopsies

SUMMARY:
The purpose of this study is the investigation of new host-microbiome interactions promoting adenoma formation and adenocarcinoma progression. For that purpose, the investigators will collect saliva, stool and colon biopsy specimens from patients referred to colonoscopy or surgical resection of colorectal tumor. Besides, a questionnaire about diet, lifestyle and medical history will be collected. Sample analysis will involve simultaneous characterization of host and microbiota genomic and transcriptomic components.

ELIGIBILITY:
Lower GI endoscopy patients

Inclusion Criteria:

* Participant is willing and able to give informed consent for the participation in the study before any protocol-specific screening procedures are performed
* Male or female, aged 18 years or above
* Referred to lower GI endoscopy. Referral reasons can be among others:

  * Positive FOBT (Fecal Occult Blood Test)
  * Follow up after polypectomy
  * Screening because of age
  * Bleeding
  * Abdominal pain
  * Familial or past history of colon cancer or adenoma
  * Abnormal imaging such as barium enema
  * Change in bowel habits
* Both self-referrals, referrals from external GP or specialists and internal referrals can be included.

Exclusion Criteria:

* Previous diagnosis of an inflammatory bowel disease
* Previous diagnosis of intestinal polyposis syndrome

CRC patients

Inclusion criteria:

* Participant is willing and able to give informed consent for the participation in the study before any protocol-specific screening procedures are performed
* Male or female, aged 18 years or above
* Diagnosis of CRC for which resection is planned
* Both internal and external referrals from specialists can be included

Exclusion Criteria:

* Previous diagnosis of an inflammatory bowel disease
* Previous diagnosis of intestinal polyposis syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants are patients with CRC that will undergo surgical tumor resection or patients referred for lower GI endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Differential host microbiome composition and abundance in healthy, adenoma and CRC patients and its correlation to CRC risk features and host genomic and transcriptomic components. | 2 years
  Host microbiome composition and abundance data will be generated from saliva, stool and colonic biopsies with amplicon-based 16S ribosomal RNA sequencing. This data will be correlated to CRC risk factors collected in a questionnaire covering lifestyle, diet and medical history as well as host genomic and transcriptomic profiling generated by targeted gene sequencing and microarray-based gene expression profiling.

CONTACTS AND LOCATIONS:
Locations (2):
- Universitaire Ziekenhuizen Leuven, Leuven, Flemish Brabant, Belgium
- Academisch Medisch Centrum, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No